CLINICAL TRIAL: NCT05562973
Title: Safety and Tolerability of Psilocybin in Post-Traumatic Stress Disorder
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The principal investigator will be at a new institution.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00288303
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Sequence 1 (15, 20, 25) (Experimental): Psilocybin dose sequence
  Session 1: 15 mg Session 2: 20 mg Session 3: 25 mg
  Interventions: Drug: Psilocybin
- Dose Sequence 2 (20, 25, 30) (Experimental): Psilocybin dose sequence
  Session 1: 20 mg Session 2: 25 mg Session 3: 30 mg
  Interventions: Drug: Psilocybin
- Dose Sequence 3 (25, 30, 35) (Experimental): Psilocybin dose sequence
  Session 1: 25 mg Session 2: 30 mg Session 3: 35 mg
  Interventions: Drug: Psilocybin
- Dose Sequence 4 (30, 35, 40) (Experimental): Psilocybin dose sequence
  Session 1: 30 mg Session 2: 35 mg Session 3: 40 mg
  Interventions: Drug: Psilocybin
- Dose Sequence 5 (35, 40, 45) (Experimental): Psilocybin dose sequence
  Session 1: 35 mg Session 2: 40 mg Session 3: 45 mg
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive three psilocybin sessions, at least two weeks apart.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and potential efficacy of psilocybin-assisted psychotherapy to reduce post-traumatic stress disorder (PTSD) severity in a sample of individuals with PTSD.

DETAILED DESCRIPTION:
The proposed Phase I study aims to evaluate the safety, tolerability, and potential efficacy of psilocybin-assisted psychotherapy to reduce PTSD severity in a sample of individuals with PTSD. A sample of up to 30 individuals with PTSD will be recruited. All participants will receive the intervention, which will consist of three psilocybin sessions with an interval of approximately 2 weeks between each session. A 3+3 Phase I trial design will be used to evaluate a range of possible dose sequences with doses ranging from 15 mg up to 45 mg. Safety, tolerability, and efficacy endpoints will be evaluated 2 weeks following each psilocybin session and at 1-month, 3-month, and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old. Participants up to 80 years old who otherwise meet safety criteria will be included to ensure generalizability to the broader clinical population of people with PTSD. Prior work (Griffiths et al. 2016) by our research team administering psilocybin to older cancer patients using the same upper age limit in the inclusion/exclusion criteria (i.e., 80 years old) found a comparable risk profile for psilocybin to research conducted with younger patients. Although it is possible that older patients experience diminished serotonin 2A (5-HT2A) receptor expression resulting in a lower/less intense response to psilocybin, this information will be important to gather in this Phase I context.
* Have given written informed consent
* Read, write, and speak English
* At Screening, meet Diagnostic and Statistical Manual-5th edition (DSM-5) criteria for current PTSD with a symptom duration of 6 months or longer according to the Clinician-Administered PTSD Scale for DSM-5
* Able to complete the study measures
* Previously sought treatment for PTSD (e.g., prolonged exposure therapy, cognitive processing therapy, sertraline, paroxetine)
* Be otherwise medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests (Complete Blood Count, Comprehensive Metabolic Panel, urine beta-human chorionic gonadotropin, urine toxicology screen).

Exclusion Criteria:

* Current physical dependence (as evidenced by self-reported withdrawal symptoms) on a drug other than caffeine or nicotine
* Seizure disorder
* Receiving current treatment for PTSD
* Cardiovascular conditions: angina, a clinically significant ECG abnormality (e.g. atrial fibrillation or corrected QT interval >450msec), transient ischemic attack (TIA) in the last 6 months, stroke, or uncontrolled hypertension with resting blood pressure systolic >150 or diastolic >95.
* Recent (<1year) intracranial or subarachnoid hemorrhage, ischemic stroke, TIA
* Pulmonary disease: chronic obstructive pulmonary disease, active asthma (inhaler use in last 6 months)
* Diabetes mellitus treated with insulin or oral hypoglycemic agents
* Current suicidal ideation or suicidality
* Current engagement in evidence-based PTSD therapy/treatment (prior to psilocybin session)
* Women: Pregnancy (pregnancy tests will be conducted for women during screen and prior to experimental sessions).
* Current or past history of meeting DSM-5 criteria for Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder.
* Currently taking efavirenz or serotonin-acting dietary supplements (e.g., 5-hydroxy- tryptophan, St. John's wort).
* Currently taking antidepressants of any drug class, antipsychotics, or monoamine oxidase inhibitors.
* Recent (within past 12 months) or extensive history of hallucinogen use (>20 lifetime uses).
* Moderate or severe DSM-5 Substance Use Disorder in the past five years (excluding tobacco and caffeine)
* Family (i.e., 1st degree relative) history of Schizophrenia, Psychotic Disorder (unless substance-induced or due to a medical condition), or Bipolar I Disorder.
* For the final (5th) dose sequence (35, 40, and 45 mg) participants that weigh less than 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Peak Post-Administration Blood Pressure | Approximately 1.5 - 2 months
  Blood pressure will be monitored at 30, 60, 90, 120, 180, 240, 300, and 360 minutes after capsule administration. Mean peak blood pressure across the 3 psilocybin sessions will be used as the outcome measure.
Mean Peak Post-Administration Heart Rate | Approximately 1.5 - 2 months
  Heart rate will be monitored at 30, 60, 90, 120, 180, 240, 300, and 360 minutes after capsule administration. The mean peak heart rate across the 3 psilocybin sessions will be used as the outcome measure.
Mean Pre-Administration Suicide Ideation Scores (Columbia Suicide Severity Rating Scale - Severity Factor) | Approximately 3 weeks
  The Columbia Suicide Severity Rating Scale will be used to assess baseline severity of suicide ideation. Scores on the Severity subscale range from 1 - 5, where 1= "wish to be dead"; 2 = "nonspecific active suicidal thoughts"; 3 = "suicidal thoughts with methods"; 4 = "suicidal intent"; and 5 = "suicidal intent with plan". The mean of the Severity subscale scores from the 3 preparation visits will be used as the outcome measure.
Mean Change in Suicide Ideation Scores (Columbia Suicide Severity Rating Scale - Severity Factor) | Approximately 3 weeks pre-administration; approximately 1.5 - 2 months post-administration
  The Columbia Suicide Severity Rating Scale will be used to assess post-administration severity of suicide ideation. Scores on the Severity subscale range from 1 - 5, where 1= "wish to be dead"; 2 = "nonspecific active suicidal thoughts"; 3 = "suicidal thoughts with methods"; 4 = "suicidal intent"; and 5 = "suicidal intent with plan". The mean change in Severity subscale scores between the preparation visits and the integration visits will be used as the outcome measure.

SECONDARY OUTCOMES:
Mean Change in Clinician-Administered PTSD Scale for DSM-5 scores | Approximately 3 weeks pre-administration; approximately 1.5 - 2 months post-administration
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a semi-structured interview that assesses history of DSM-5-defined traumatic event exposure, including the most distressing event, time since exposure, to produce a diagnostic score (presence vs. absence) and a PTSD Total Severity score. The mean of the Total Severity scores from the 3 integration visits will be used as the outcome measure.
Mean Change in PTSD Checklist Scores | Approximately 3 weeks pre-administration; approximately 1.5 - 2 months post-administration
  The PTSD Checklist (PCL-5) is a 20-item self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms according to diagnostics in the DSM-5. Participants indicate how much distress they have experienced due to symptoms such as "Trouble remembering important parts of a stressful experience from the past" and "Feeling irritable or having angry outbursts" on a five-point Likert-type scale (1=Not at all to 5=Extremely). The mean of the PCL-5 scores from the 3 integration visits will be used as the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Johnson, Ph.D., Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165